CLINICAL TRIAL: NCT06199830
Title: A Case-control Study on the Differentiation Between Cough Variant Asthma and Chronic Cough
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-KLS-100-01
Record Dates: First submitted 2023-10-20; First posted 2024-01-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-12

CONDITIONS: Asthma
Keywords: small airway dysfunction; cough variant asthma; Chronic cough
MeSH Terms: conditions — Asthma; Cough-Variant Asthma; Chronic Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- cough variant asthma: (1) chronic cough (≥8 weeks) as the sore or predominant symptom; (2) variable airway limitation evaluated by BHR test; (3) a positive response to anti-asthma therapy; (4) No other causes of chronic cough.
  Interventions: Diagnostic Test: positive bronchial provocation test
- chronic cough: (1) chronic cough (≥8 weeks) as the sore or predominant symptom; (2) without radiographic evidence of lung disease; (3) with no fever, blood-stained sputum or other active respiratory injection;

INTERVENTIONS:
Diagnostic Test: positive bronchial provocation test — Patients were asked to inhale gradually increasing doses of methacholine (0.9% saline, 0.078, 0.312, 1.125 and 2.504 mg), and FEV1 was measured after each inhalation. This test was stopped until a reducing in baseline FEV1 of 20%.
  Groups: cough variant asthma

SUMMARY:
this study aimed to compare characters in pulmonary function of patients with cough variant asthma and chronic cough and establish a diagnostic model.

DETAILED DESCRIPTION:
the investigators retrospectively collected information from patients with chronic cough who underwent pulmonary tests at the First Affiliated Hospital of Zhejiang Chinese Medical University from January 2019 to December 2019. Data of external test were also from the First Affiliated Hospital of Zhejiang Chinese Medical University, and time period was from January 2023 to April 2023.Pulmonary function test and methacholine challenge test was performed by professional technicians. Characters between patients with cough variant asthma and chronic cough were compared to establish a diagnostic model.

ELIGIBILITY:
Inclusion Criteria:

* (1) age from 18 years old to 65 years old; (2) clinical diagnosis of CVA and CC .

Exclusion Criteria:

* Exclusion criteria for CVA were: a history of COPD, bronchiectasis, bronchitis, cystic fibrosisor pneumonia, interstitial lung disease, pulmonary tuberculosis, lung cancer; cough caused by drugs or treatments; patients with upper airway cough syndromes (UACS) and gastroesophageal reflux-related cough (GERC) or other apparent causes of cough; patients who used corticosteroid (ICS) in the previous four weeks; Exclusion criteria for CC were: a history of variable airway limitation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospectively collected information from patients with CC who underwent pulmonary tests at the First Affiliated Hospital of Zhejiang Chinese Medical University from January 2019 to December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
positive bronchial provocation test | up to 1 week
  Patients were asked to inhale gradually increasing doses of methacholine (0.9% saline, 0.078, 0.312, 1.125 and 2.504 mg), and FEV1 was measured after each inhalation. This test was stopped until a reducing in baseline FEV1 of 20%

SECONDARY OUTCOMES:
small airway dysfuction | up to 1 week
  MMEF% pred, FEF50% pred, FEF75% pred

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Yang, Dr, Principal Investigator — The First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, China

REFERENCES:
- [Derived] Ni K, Wang S, Zhang X, Liu S, Zhang Y, Li Y, Wang Y, Yang J. Association between clinical and pulmonary function features and diagnosis of cough variant asthma: a case-control study. BMJ Open. 2025 Feb 22;15(2):e084721. doi: 10.1136/bmjopen-2024-084721. PMID 39987008